CLINICAL TRIAL: NCT04160910
Title: 5HTP Regulation Of Asthma In Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kirsten Kloepfer, Assistant Professor of Pediatrics; Division of Pulmonary, Allergy and Sleep Medicine; Riley Hospital for Children at Indiana University Health, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Kloepfer_1902366300
Record Dates: First submitted 2019-10-24; First posted 2019-11-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Mild or Moderate Asthma With Allergic Sensitization
MeSH Terms: conditions — Lymphoma, Follicular | interventions — 5-Hydroxytryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 5-hydroxytryptophan (Active Comparator): Dosage of 5-hydroxytryptophan will be determined by weight:
  If subject weighs less than 100lbs: 50mg twice a day If subject weights more than 100lbs: 100mg twice a day
  Interventions: Drug: 5-Hydroxytryptophan
- Placebo (Placebo Comparator): Dosage of placebo will be determined by weight:
  If subject weighs less than 100lbs: 50mg twice a day If subject weights more than 100lbs: 100mg twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-Hydroxytryptophan — Double blinded placebo controlled. 28 day dosing period followed by 3 week washout period. Then crossover to other arm of study
  Other Names: 5HTP
  Arms: 5-hydroxytryptophan
Drug: Placebo — Double blinded placebo controlled. 28 day dosing period followed by 3 week washout period. Then crossover to other arm of study
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about if taking a supplement called 5-hydroxytryptophan (5HTP) can improve breathing and anxiety symptoms related to asthma. To help learn more subjects will either be assigned to a group that is taking the supplement (5HTP) or a group that is taking a placebo. This will be decided randomly. Later in the study subjects will crossover to the other group.There are 5 study visits over the course of about 12 weeks.

DETAILED DESCRIPTION:
The objective of this study is to test the hypothesis that over-the-counter amino acid supplement 5HTP (isolated from the plant Griffonia Simplifolia) reduces human allergic lung responses and consequently improves lung function. The primary outcome is the change in FEV1. We anticipate the 5HTP at the proposed doses will improve lung function as in preclinical studies that used clinically relevant 5HTP. Secondary outcomes will be blood eosinophil counts and reduced symptoms for anxiety/depression, as seen in changes in the anxiety-depression scores from questionnaires (CES-DC & SCARED). The results from these studies have the transformative potential to influence approaches to improve lung function and asthma-associated anxiety/depression.

* Aim 1: Test that 5HTP improves lung function in children with allergic asthma
* Aim 2: Test that 5HTP reduces eosinophil numbers in the blood and nasal fluid of patients with asthma from Aim 1
* Aim 3: Test that 5HTP decreases lung inflammation, increases cortisol and prolactin without altering systemic plasma concentrations of 5HTP, serotonin, 5-hydroxyindoleacetic acid (5-HIAA), and dopamine

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 Years of Age
* Mild to Moderate Asthma based on ATS guidelines
* Positive Allergy Test (positive skin or serum IgE)
* Weight ≥ 70 lbs (32 kg)
* CES-DC cut-off ≥ 15 (total score range is 0 to 60) or SCARED cut-off

  * 25 (total score range is 0 to 142)
* Ability to comply with study visits and study procedures
* Informed Consent by participant and if applicable the parent or legal guardian

Exclusion Criteria:

* Currently taking a SSRI
* Taking a leukotriene inhibitor (montelukast, Zileuton)
* Severe Asthma Based on ATS Guidelines
* Taking a biologic medication (omalizumab, mepolizumab, benralizumab, dupilumab)
* Medical History of Adverse Reaction to 5HTP
* Physical findings that would compromise the safety of the study or the quality of the study data

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Testing will be performed to assess for a change in Forced Expiratory Volume at one second (FEV1) | 77 days
  Pulmonary function testing will be performed at Baseline, Day 28, and Day 49, and Day 77

SECONDARY OUTCOMES:
Blood will be obtained to assess Eosinophil Count | 77 days
  Will be performed at Baseline, Day 28, and Day 49, and Day 77
Questionnaires will be utilized to look for a decrease in symptoms for Anxiety/Depression Reduced Symptoms for Anxiety/Depression | 77 days
  Changes in Anxiety/Depression will be determined via questionnaire that will be administered at Baseline, Day 28, and Day 49, and Day 77 . Will use the Center for Epidemiological Studies Depression Scale for Children (CES-DC) to measure depression and Screen for Child Anxiety Related Disorders (SCARED)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Kloepfer, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No